CLINICAL TRIAL: NCT03665506
Title: A Non-interventional Study to Assess Effectiveness and Safety of Trifluridin/tipiracil in Patients with Metastatic Colorectal Cancer
Brief Title: Trifluridin/tipirACil in MeTastatIc Colorectal Cancer
Acronym: TACTIC
Status: Completed | Type: Observational
Sponsor: Servier (Industry)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-040380
Record Dates: First submitted 2018-08-26; First posted 2018-09-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; Trifluridin/Tipiracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Trifluridin/Tipiracil — QoL assessment
  Other Names: QoL assessment

SUMMARY:
A non-interventional, prospective, open, multicenter study in Germany in patients with metastatic colorectal cancer who have been previously treated with, or are not considered candidates for, available therapies and with decision for treatment with trifluridin/tipiracil.

DETAILED DESCRIPTION:
The purpose of this NIS, after market approval of trifluridin/tipiracil as treatment for mCRC patients who have been previously treated with, or are not considered candidates for, available therapies, is to evaluate effectiveness, QoL, treatment details and safety of trifluridin/tipiracil treatment in a real-world setting. In addition, therapy management and health economic parameters regarding trifluridin/tipiracil treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Patients with mCRC who have been previously treated with, or are not considered candidates for, available therapies including fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapies, anti-VEGF agents, and anti-EGFR agents.
* Indication for treatment as assessed by the treating physician.
* Decision for treatment with trifluridin/tipiracil.
* Signed written informed consent.
* Criteria according to current Summary of Product Characteristics (SmPC) for patients treated with trifluridin/tipiracil.
* Ability to read and understand German.

Exclusion Criteria:

* Contraindications according to SmPC for metastatic colorectal cancer patients treated with trifluridin/tipiracil.
* Participation in a clinical trial within 30 days prior to enrollment or simultaneous participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic colorectal cancer (mCRC) who have been previously treated with, or are not considered candidates for, available therapies including fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapies, anti-VEGF (vascular endothelial growth factor) agents, and anti-EGFR (epidermal growth factor receptor) agents and with decision for treatment with trifluridin/tipiracil.
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | Baseline up to 3 years
  time from first administration of trifluridin/tipiracil to death from any cause

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to 3 years
  PFS: time from first administration of trifluridin/tipiracil to disease progression or death from any cause
Overall response rate | Baseline up to 3 years
  ORR: the proportion of patients whose best response was a complete or partial response
Disease control rate 8 weeks | Baseline up to 3 years
  DCR-8: the proportion of patients with a best response of complete or partial response or stable disease, with the assessment of stable disease made at least 8 weeks after first administration of trifluridin/tipiracil
Trifluridin/tipiracil treatment details | Baseline
  Line of Trifluridin/Tipiracil treatment (Descriptive statistics using frequency tables will be used to assess the number of prior palliative systemic antineoplastic treatment regimen)
Trifluridin/tipiracil treatment details | Baseline up to 3 years
  Treatment duration
Trifluridin/tipiracil treatment details | Baseline up to 3 years
  Dose intensity (absolute and relative)
Trifluridin/tipiracil treatment details | Baseline up to 3 years
  Treatment sequence (previous and subsequent therapies in relation to Trifluridin/Tipiracil treatment) (Descriptive statistics using frequency tables will be used to assess previous and subsequent palliative systemic antineoplastic treatment regimen used.)
AEs and SAEs according to NCI CTCAE | Baseline up to 3 years
  AEs and SAEs according to NCI CTCAE
Safety laboratory values of participants | Baseline up to 3 years
  By-patient display of all safety laboratory results captured as per clinical routine (e.g. CEA, CA 19-9, haemoglobin, neutrophils absolute, lymphocytes count, platelets count, leukocytes count, alkaline phosphatase, ALT (GPT), AST (GOT), bilirubin total and serum creatinine). In addition, CTCAE grades of neutrophils, white blood cell count, platelets, haemoglobin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, alkaline phosphatase and creatinine will be presented using frequencies and percentages for each visit. Shift tables opposing CTCAE grades during treatment to baseline CTCAE grades of the mentioned parameters will also be presented per visit using frequencies and percentages.
Therapy management (use of relevant supportive medications) | Baseline up to 3 years
  Number of patients receiving G-CSFs for prophylaxis of chemotherapy-induced neutropenia and febrile neutropenia (Frequencies)
Patient-reported outcomes (PROs) on quality of life (QoL) | Baseline up to 3 years
  PRO-CTCAE: Questionnaire PRO-CTCAE is used to determine patients' symptomatic toxicity. Item cluster scores of PRO-CTCAE questionnaire at each visit and change from baseline of scores.
Patient-reported outcomes (PROs) on quality of life (QoL) | Baseline up to 3 years
  EQ-5D-5L: Questionnaire EQ-5D-5L is used to determine patients' health related quality of life. EQ-5D-5L index and visual analogue score at each visit and change from baseline for both, index and visual analogue score.

OTHER OUTCOMES:
Time to deterioration of the ECOG performance status | Baseline up to 3 years
Assessment of health economic parameters | Baseline up to 3 years
  Incidence of hospitalization (Frequencies)
Assessment of health economic parameters | Baseline up to 3 years
  Frequency of hospitalization (Frequencies)
Assessment of health economic parameters | Baseline up to 3 years
  Total duration of hospital stays per patient (descriptive statistics)
Assessment of health economic parameters | Baseline up to 3 years
  Reasons for hospitalizations per patient and per case (Frequencies)
Assessment of health economic parameters | Baseline up to 3 years
  Number of consultations of various medical specialists
Assessment of health economic parameters | Baseline up to 3 years
  Incidence of home care (Frequencies)
Assessment of health economic parameters | Baseline up to 3 years
  Location of terminal care (Frequencies)

CONTACTS AND LOCATIONS:
Locations (1):
- Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kroning H, Gohler T, Decker T, Grundeis M, Kojouharoff G, Lipke J, Semsek D, Moorahrend E, Sauer A, Bruch HR, Liersch R, Nusch A, Vehling-Kaiser U, Welslau M, Grunewald R, Harich HD, Stephany M, Uhlig J, de Buhr R, Frank M, Hogrefe C, Marschner N, Potthoff K, Hartmann F, Reislander T, Schwaner I. Effectiveness, safety and quality of life of trifluridine/tipiracil in pretreated patients with metastatic colorectal cancer: Real-world data from the noninterventional TACTIC study in Germany. Int J Cancer. 2023 Sep 15;153(6):1227-1240. doi: 10.1002/ijc.34603. Epub 2023 Jun 1. PMID 37260368